CLINICAL TRIAL: NCT02306993
Title: Sickle Cell Hemoglobinopathies and Bone Heath
Brief Title: Sickle Cell Hemoglobinopathies and Bone Health
Status: Active, not recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Biree Andemariam, Professor, UConn Health
Other Study IDs: 14-136-6
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Sickle Cell Trait
Keywords: Sickle Cell Disease (SCD); Sickle Cell Trait (SCT)
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be collected once from each subject by certified study staff at UCHC, CCMC or the participating approved community sites in a private setting.Subjects will donate ~12-15 cc of whole blood via venipuncture. Blood will be collected into 3 vacutainer tubes: one 3.5-mL lavender top tube for CBC and hemoglobin electrophoresis, one 3.5-mL yellow top tube for serum calcium and phosphate, and one 5-mL red-top tube for 25-OH vitamin D, P1NP, CTX, and PTH analysis. The
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy volunteers without SCT: Includes Healthy African American female volunteer between the ages of 18 and 45 years without sickle cell trait. Their blood and bone density x-ray will help researchers gain a better understanding of what might be different about the way having sickle cell trait affects bone.
  Interventions: Other: Healthy volunteers without SCT
- Healthy volunteers with SCT: Includes Healthy African American female volunteer between the ages of 18 and 45 years with sickle cell trait. Their blood and bone density x-ray will help researchers gain a better understanding of what might be different about the way having sickle cell trait affects bone.
  Interventions: Other: Healthy volunteers with SCT
- Volunteers with SCD: Healthy African American female volunteer between the ages of 18 and 45 years with sickle cell disease. Their blood and bone density x-ray will help researchers gain a better understanding of what might be different about the way having sickle cell disease affects bone.
  Interventions: Other: Volunteers with SCD

INTERVENTIONS:
Other: Healthy volunteers without SCT — Subjects will undergo bone density evaluation via dual energy x-ray absorptiometry (DEXA) scanning. Subjects will provide a sample of for testing of bone turnover markers, complete blood count, and hemoglobin electrophoresis. Subjects will provide information about their dietary calcium intake and pain burden.
  Groups: Healthy volunteers without SCT
Other: Healthy volunteers with SCT — Subjects will undergo bone density evaluation via dual energy x-ray absorptiometry (DEXA) scanning. Subjects will provide a sample of for testing of bone turnover markers, complete blood count, and hemoglobin electrophoresis. Subjects will provide information about their dietary calcium intake and pain burden.
  Groups: Healthy volunteers with SCT
Other: Volunteers with SCD — Subjects will undergo bone density evaluation via dual energy x-ray absorptiometry (DEXA) scanning. Subjects will provide a sample of for testing of bone turnover markers, complete blood count, and hemoglobin electrophoresis. Subjects will provide information about their dietary calcium intake and pain burden.
  Groups: Volunteers with SCD

SUMMARY:
This research study has two purposes. The first purpose is to determine whether having sickle cell trait (SCT) is a risk factor for the development of bone thinning at an earlier age than expected. Nearly 10% of African Americans (AA) carry sickle cell trait and most of them are unaware of it. African Americans are less likely to develop thin bones than whites, but if they sustain a bone fracture, they are more likely to die from it. We believe having sickle cell trait may lead to bone thinning and predispose a subset of African Americans to dangerously thin bones. The second purpose is to try to understand why individuals with sickle cell disease (SCD) have thinner bones than healthy individuals do. Doctors have already discovered that people with sickle cell disease have very thin bones, but they have not determined why. Our study will try to identify whether the bone thinning is from the body not making enough bone or from the body losing bone once it is made.

DETAILED DESCRIPTION:
SCD is a hereditary disease arising only when two parents carrying sickle cell trait (SCT) conceive a child. SCT is clinically silent but very common in African Americans with a ~10% prevalence, although most carriers are unaware of their status. There are no data on bone mineral density (BMD) or vitamin D status in these individuals. Although it is clear that those with SCD have accelerated bone thinning the effect of SCT on bone metabolism or fractures has not been studied. Although the incidence of hip fracture in AA women is about half that of white women, the etiology and risk factors of fractures in AA women are not clearly defined, and it is intriguing to postulate that SCT may have a relationship to bone metabolism and fracture risk in this population, and thus contribute to racial disparity. We hypothesize that the mechanisms underlying altered bone homeostasis in SCD are different than in the general population but perhaps similar to those with SCT. We also hypothesize that SCT is a state of reduced bone mineralization which may contribute to racially disparate outcomes among AAs with bone fractures. Our objectives are (1) to define the mechanisms of bone loss in SCD and (2) to evaluate parameters of bone metabolism in human subjects with SCT compared to those with normal hemoglobin and those with SCD. We will investigate the effect of SCD and SCT on bone homeostasis in premenopausal AA subjects via serum bone turnover markers, calciotrophic hormones and bone mineral density (BMD) testing. We hypothesize that premenopausal AA women with SCT will have significantly lower BMD and higher serum bone turnover markers than race- and age-matched control AA women. In addition, we will explore Vitamin D status and its relationship to bone turnover and BMD in all three groups. We further postulate that bone homeostasis in SCT subjects will be intermediate between healthy controls and subjects with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years.
* Female.
* Regular menstrual periods.
* Self-identification of African American race.

Exclusion Criteria:

* Taking oral contraceptives or medications known to influence bone metabolism (e.g. Glucocorticoids, anti-resorptive or anabolic medications for osteoporosis, pharmacologic Vit D dosing).
* Known metabolic bone disorder (e.g. uncontrolled thyroid disease, hyperparathyroidism).
* Pregnant, breast-feeding, or within 3 months post-partum.
* Taking an investigational drug.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population includes healthy African American female volunteers with and without SCT and African American female volunteers with SCD.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin genotype with serum bone turnover markers and bone density | 3 years
  Assess the association of hemoglobin genotype with serum bone turnover markers and bone density.

CONTACTS AND LOCATIONS:
Overall Officials: Biree Andemariam, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States